CLINICAL TRIAL: NCT00283374
Title: A Prospective, Longitudinal Multicenter, Nontreatment, Exploratory Biomarker Study of Metabolic Syndrome in Subjects Undergoing Laparoscopic Roux-En-Y Gastric Bypass Bariatric Syndrome
Brief Title: Study Evaluating Metabolic Syndrome in Subjects Undergoing Gastric Bypass Bariatric Syndrome
Status: Terminated | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 9804Z1-900
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-05

CONDITIONS: Morbid Obesity; Metabolic Disease
Keywords: Metabolic Syndrome; Obesity; Nonalcoholic fatty liver disease; Nonalcoholic steatohepatitis; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid; Metabolic Diseases; Metabolic Syndrome; Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-Y Gastric Bypass

SUMMARY:
Metabolic syndrome is rapidly emerging as an epidemic of global proportions and its definition is still evolving. Patients with this syndrome are at increased risk for cardiovascular disease, and at increased risk of mortality from cardiovascular disease.

Metabolic syndrome is strongly associated with obesity, and more specifically with abdominal obesity. Abdominal obesity, comprises two main components: visceral (VAT) and subcutaneous (SAT) adipose tissue depots, with VAT reported as more metabolically active than SAT, and thought to play a major role in the metabolic disturbances associated with obesity and metabolic syndrome.

Non-alcoholic fatty liver disease (NAFLD) is fast becoming the most common liver disease and is associated with obesity, insulin resistance and metabolic syndrome.

Bariatric surgery has yielded dramatic results including longitudinal loss of excess body weight and either complete reversal or significant improvement of several features of metabolic syndrome, NAFLD, and nonalcoholic steatohepatitis (NASH) in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be approved by both insurance and site standard of care to undergo the Roux-en-Y gastric bypass procedure
* Male and Female Candidates for Roux-en-Y Bariatric Surgery
* Must be diagnosed with Metabolic Syndrome; having abdominal obesity and at least 2 other features of the syndrome per IDF (International Diabetes Foundation)
* Obese control group:Subjects should be obese and should not have any other features of metabolic syndrome.

Exclusion Criteria:

* Any subjects with prior bariatric surgery
* No other major surgery within the last 6 months
* Diabetes on treatment with hypoglycemic medication in the previous 6 months

Other exclusions apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Italy, decresg@wyeth.com; Trial Manager, Principal Investigator — For Sweden, MedInfoNord@wyeth.com
Locations (14):
- United States (9):
  - Irvine, California
  - Orange, California
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
- Italy (3):
  - Aosta
  - Pisa
  - Roma
- Sweden (2):
  - Gothenburg
  - Stockholm